CLINICAL TRIAL: NCT00387517
Title: An Eight-week Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren / HCTZ (150/25 mg and 300/25 mg) in Comparison With HCTZ 25 mg in Patients With Essential Hypertension Not Adequately Responsive to HCTZ 25 mg Monotherapy
Brief Title: Safety/Efficacy of Combo Therapy With Aliskiren & Hydrochlorothiazide vs Therapy With Hydrochlorothiazide Alone in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2333
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Diastolic; systolic; hypertension; aliskiren; blood pressure; hydrochlorothiazide; HCTZ
MeSH Terms: conditions — Hypertension; Heart Murmurs; Systolic Murmurs

INTERVENTIONS:
Drug: Aliskiren/HCTZ

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of combination therapy of aliskiren/hydrochlorothiazide (HCTZ) 150/25 mg and 300/25 mg compared with HCTZ 25 mg in patients with hypertension who do not show response to HCTZ 25 mg over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years old or older.
* Patients with a diagnosis of hypertension defined as follows:

  * Newly diagnosed patients or patients who have not been treated for hypertension within the 4 weeks prior to Visit 1 must have a msDBP >= mmHg and < 110 mmHg at Visit 1.
  * All patients who have been treated for hypertension within the 4 weeks prior to Visit 1 must have a msDBP >= 85 mmHg and < 110 mmHg at Visit 2.
  * All patients must have a msDBP >= 90 mmHg and < 110 mmHg at Visit 5.
* Patients who are eligible and consent to participate in the study

Exclusion Criteria:

* Severe hypertension (msDBP >= 110 mmHg and/or MSSBP >=180 mmHg).
* Previous or current diagnosis of heart failure.
* History of hypertensive encephalopathy or cerebrovascular accident, transient ischemic cerebral attack, myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean sitting diastolic blood pressure lowering effect at baseline, and week 8.

SECONDARY OUTCOMES:
Mean sitting systolic blood pressure (msDBP) lowering from baseline to week 8
Safety and tolerability
Proportion of patients achieving a blood pressure control target at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Blumenstein M, Romaszko J, Calderon A, Andersen K, Ibram G, Liu Z, Zhang J. Antihypertensive efficacy and tolerability of aliskiren/hydrochlorothiazide (HCT) single-pill combinations in patients who are non-responsive to HCT 25 mg alone. Curr Med Res Opin. 2009 Apr;25(4):903-10. doi: 10.1185/03007990902804158. PMID 19245300